CLINICAL TRIAL: NCT05797818
Title: The Effect of Red Light Photobiomodulation and Topical Disinfectants on the Nasal Microbiome
Brief Title: Red Light Photobiomodulation and Topical Disinfectants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ondine Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 31686-2022
Record Dates: First submitted 2023-01-26; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-02

CONDITIONS: Healthcare Associated Infection; Nosocomial Infection; Surgical Site Infection
Keywords: Staphylococcal aureus; Methylene blue; Chlorhexidine gluconate; Nasal decolonization; Photobiomodulation; Photodynamic therapy; Nasal microbiome
MeSH Terms: conditions — Cross Infection; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: A single open-label healthy group is being evaluated for any changes to the normal nasal microbiome. Each week nasal cultures will be done and the subject exposed to different interventions including red light alone, and several disinfectants. Nasal cultures will be done for 48 hours after the intervention to determine the effect, if any, on the nasal microbiome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Methylene Blue (Experimental): All subjects will have an initial baseline culture done of their nasal microbiome followed by an administration of 0.01% methylene blue solution. Next, subjects will undergo two minute of non-thermal red light exposure. A second round of solution administration and light exposure will be repeated resulting in 4 minutes of red light exposure.
  Once the treatment has been completed, a new culture will be taken from the subjects nares followed by one at 4-, 8-, 24-, and 48-hours after treatment.
  Interventions: Device: Methylene Blue Only
- Chlorhexidine gluconate (Experimental): All subjects will have an initial baseline culture done of their nasal microbiome followed by an administration of 0.25% chlorhexidine solution. Next, subjects will undergo two minute of non-thermal red light exposure. A second round of solution administration and light exposure will be repeated resulting in 4 minutes of red light exposure.
  Once the treatment has been completed, a new culture will be taken from the subjects nares followed by one at 4-, 8-, 24-, and 48-hours after treatment.
  Interventions: Device: Chlorhexidine Gluconate Only
- Methylene blue and Chlorhexidine gluconate (Experimental): All subjects will have an initial baseline culture done of their nasal microbiome followed by an administration of 0.01% methylene blue and 0.25% chlorhexidine gluconate solution. Next, subjects will undergo two minute of non-thermal red light exposure. A second round of solution administration and light exposure will be repeated resulting in 4 minutes of red light exposure.
  Once the treatment has been completed, a new culture will be taken from the subjects nares followed by one at 4-, 8-, 24-, and 48-hours after treatment.
  Interventions: Device: Methylene Blue + Chlorhexidine Gluconate
- Light Only (Experimental): All subjects will have an initial baseline culture done of their nasal microbiome followed by 4 minutes of non-thermal red light exposure.
  Once the treatment has been completed, a new culture will be taken from the subjects nares followed by one at 4-, 8-, 24-, and 48-hours after treatment.
  Interventions: Device: Light Only

INTERVENTIONS:
Device: Methylene Blue Only — All subjects will have a baseline sample taken of their nasal microbiome and undergo the administration of the following:
  - Methylene Blue (0.01%) + 4 minutes of light treatment
  Arms: Methylene Blue
Device: Chlorhexidine Gluconate Only — All subjects will have a baseline sample taken of their nasal microbiome and undergo the administration of the following:
  - Chlorhexidine gluconate (0.25%) + 4 minutes of light treatment
  Arms: Chlorhexidine gluconate
Device: Methylene Blue + Chlorhexidine Gluconate — All subjects will have a baseline sample taken of their nasal microbiome and undergo the administration of the following:
  - Methylene blue (0.01%) + chlorhexidine gluconate (0.25%) + 4 minutes of light treatment
  Arms: Methylene blue and Chlorhexidine gluconate
Device: Light Only — All subjects will have a baseline sample taken of their nasal microbiome and undergo the administration of the following:
  - 4 minutes of light treatment only
  Arms: Light Only

SUMMARY:
The goal of this clinical trial is to evaluate the potential effects of photobiomodulation when used with topical disinfectants in the anterior nares of healthy adults.

Over a three week period, participants will have their anterior nares swabbed with methylene blue, chlorhexidine gluconate, or a combination of the two followed by 4 minutes of non-thermal red light treatment. The fourth week of consist of only red light treatment. Culture samples of the subjects nasal microbiome will be taken prior to treatment, immediately after treatment, 4-, 8-, 24-, and 48 hours after treatment.

DETAILED DESCRIPTION:
This is an exploratory, single-center, open-label, single-arm study with microbiological endpoint using photobiomodulation (PBM) and topical disinfectants to determine the effect on the nasal microbiota.

The photobiomodulation system distributes about 700mW of light to each nostril using a 2-channel diode laser with non-thermal, red light. The topical disinfectants are methylene blue (0.01%) and chlorhexidine gluconate (0.25%). Following a pretreatment nasal culture, these two disinfectants will be administered into the patient's anterior nares followed by a two-minute light cycle. This process is repeated once more resulting in two treatments cycles (4-minutes total). Following this, nasal cultures are taken immediately and at 4-, 8-, 24-, and 48- hours. Broad spectrum and Staphylococcus spp. culturing of nasal swabs will be conducted. Swabs will also be submitted for Next Generation Sequencing to characterize the effect of light and disinfectants on the nasal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older

Exclusion Criteria:

* Pregnant Women
* Those Under 18 years of age
* Prisoners
* Mentally Disabled Persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Effect of PBM with Topical Disinfectants (Quantitative) | The change in bacterial bioburden during the week of each of the four weeks respective intervention.
  The Quantitative outcome measure is the change from baseline in nasal bacterial bioburden (measured in CFU/mL) by the effects of red light photobiomodulation on nasal bacteria when used with and without topical disinfectants. Each subject's baseline nasal bacterial level is determined prior to the weekly intervention. There are no subject reported outcome measures.
Effect of PBM with Topical Disinfectants (Semi-Quantitative) | The change in bacterial bioburden during the week of each of the four weeks respective intervention.
  The Semi-quantitative outcome measure is the change in bacterial growth between different time points measured by the number of quadrants with bacterial growth on a culture plate. Photographs of each culture plate will allow visual comparisons between time points. Each subject's baseline nasal bacterial level is determined prior to the weekly intervention.

SECONDARY OUTCOMES:
Effect of PBM with Topical Disinfectants (NGS) | The change in bacterial bioburden during the week of each of the four weeks respective intervention.
  Nasal culture responses over several days will be evaluated using Next Generation Sequencing (NGS) to determine how long it takes for the nasal microbiome to return to its previous non-treated level. NGS allows for determining what percentage of the total microbiome a certain species of bacteria is.

CONTACTS AND LOCATIONS:
Overall Officials: ROGER ANDERSEN, MD, MPH, Principal Investigator — Ondine Biomedical
Locations (1):
- Ondine Research Laboratories, Bothell, Washington, United States

IPD SHARING:
Plan to Share IPD: No